CLINICAL TRIAL: NCT06712264
Title: Construction and Effectiveness Evaluation of Painless Digestive Endoscopy Mode Led by Anesthesia Nurses Under the Guidance of Anesthesiologists
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jixiangyu, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYEC2024-234
Record Dates: First submitted 2024-11-24; First posted 2024-12-02 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Endoscopy, Gastrointestinal
Keywords: Painless endoscopy; Anesthesia doctors guide anesthesia nurses; sedation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Group: Sedation administered by anesthetic nurses under the guidance of anesthesiologists
- Unexposed Group: Sedation administered by anesthesiologists

SUMMARY:
The purpose is to verify the effectiveness and safety of the painless digestive endoscopy mode led by anesthesia nurses under the guidance of anesthesiologists.

DETAILED DESCRIPTION:
1. Research background Painless diagnosis and treatment, as a treatment method to alleviate patients' pain and avoid psychological and physiological adverse reactions caused by pain, has gradually expanded its application scope. With the increasing demand for comfortable healthcare in society, how to efficiently and safely implement painless diagnosis and treatment has become a focus of clinical attention. Gastrointestinal endoscopy has received increasing attention and is the gold standard for gastrointestinal examinations. WHO recommends that people over 20 years old undergo gastrointestinal endoscopy. Statistics show that in 2021, the number of gastrointestinal endoscopy examinations in China was 38 million, and it is estimated that the number of people who need to undergo gastrointestinal endoscopy examinations in China will exceed 100 million by 2030. With the improvement of living standards and the deepening of the concept of comfortable medical care, more and more people choose painless gastroscopy. The number of painless gastroscopy in China has skyrocketed since 2010. In 2005, the painless rate was less than 10%, and it gradually increased after 2010. The results of a survey on the implementation status of painless gastroscopy in China published in BJA in 2020 showed that the overall painless rate of gastroscopy in China is around 45%, and there has been great progress in the painless rate as soon as possible. However, there is a big gap between the painless diagnosis and treatment of gastroscopy in China and Europe and America, and the sedation rate of gastroscopy in Europe and America has approached 100%.

   The main problem causing this situation is the severe shortage of anesthesiologists in China at present. The current number of anesthesiologists in China is 100000, with a shortage of up to 250000 anesthesiologists. The existing number of anesthesiologists is already struggling to cope with the annual surgical workload of nearly 60 million researchers. Long term high workload and high pressure have led to a constant occurrence of overwork and death among anesthesiologists. Anesthesiology is the department with the highest sudden death rate among all clinical departments.

   In this context, researchers creatively proposed and implemented a painless diagnosis and treatment model led by anesthesia nurses under the guidance of anesthesiologists in 2019, which improved work efficiency and economic resource utilization, saved medical costs, met the people's demand for comfortable diagnosis and treatment, and effectively solved the problem of shortage of anesthesiologists. However, there is still a lack of unified standards for the training, assessment, admission, supervision, and diagnosis and treatment processes of anesthesia nurses involved in the effective operation of this model, and its effectiveness and safety also lack convincing evidence.
2. Research objective Verify the effectiveness and safety of the painless digestive endoscopy mode led by anesthesia nurses under the guidance of anesthesiologists.
3. Research significance Through this study, we will further standardize the training, assessment, admission, supervision, and diagnosis and treatment processes for anesthesia nurses, and verify the effectiveness and safety of this model through quality evaluation tools and indicators such as doctor-patient satisfaction. This will provide a basis for the further promotion of this model and open up a new path for the effective development of comfortable medical safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years old,
* no oral intake before surgery: liquid for 2 hours, solid for 6 hours.

Exclusion Criteria:

* American Society of Anesthesiology (ASA) classification greater than III,
* sleep apnea,
* allergies to soybeans, eggs, or peanuts,
* pregnancy,
* previous anesthesia related complications,,
* potential difficult ventilation,
* acute gastrointestinal bleeding,
* sub intestinal obstruction,
* severe chronic obstructive pulmonary disease (COPD)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population undergoing gastrointestinal endoscopy examination at Qingdao University Affiliated Hospital from December 2024 to February 2025.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Sedation related adverse events | During the anesthesia process
  During and after the examination process summarized by the adverse event reporting tool, the incidence of adverse events such as hypotension, hypertension, tachycardia, bradycardia, arrhythmia, hypoxemia, apnea, coughing (continuous coughing without wheezing, considered as a single cough), and body movements (non directive limb movements) were recorded. The incidence of adverse events during painless endoscopic diagnosis and treatment by anesthesiologists and anesthesiologists, as well as the number and reasons for anesthesiologists seeking help from anesthesiologists, were also recorded

SECONDARY OUTCOMES:
Patient satisfaction | During surgery
  Complete a Patient Satisfaction Survey (PSSI) before the patient leaves the hospital, using a 100mm Visual Analog Scale (VAS) (0=completely dissatisfied, 100=completely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China